CLINICAL TRIAL: NCT05167617
Title: Vitamin D Supplemental Therapy for Asthmatic Children May Improve Clinical Manifestations and Reduce IgE Serum Levels
Brief Title: Vitamin D Improves Clinical Manifestations in Asthmatic Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed B.Hamza, Clinical Professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 34960/10/21
Record Dates: First submitted 2021-11-21; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin Deficiency (Experimental)
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Vit D — Vit D was provided as 2000 IU daily for 3 and 6 months for patients who had mild and moderate HVD, respectively.

SUMMARY:
Objectives: Evaluation of the effect of vitamin D supplemental therapy (VDST) on clinical manifestation of bronchial asthma (BA) as judged by The International Study of Asthma and Allergies in Childhood (ISAAC) questionnaire and estimated serum levels of immunoglobulin E (IgE).

Patients & Methods: scores of ISAAC questionnaire and blood samples were obtained for estimation of serum IgE and 25-hydroxy VD (25-HVD) at booking time (T1) of 102 BA patients. VDST was provided as 2000 IU daily for 3 and 6 months for patients had moderate and mild HVD, respectively. At the end of 12-m after start of VDST (T2), ISAAC questionnaire and serum levels of 25-HVD and IgE were re-evaluated and the percentage of change was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age group of 6-14 years, free of exclusion criteria and complaining of chest wheezes were included in the study.

Exclusion Criteria:

* Presence of acute asthmatic attack, current or recurrent chest infection, allergic dermatological disorders, chronic rhino-sinusitis, deviated nasal septum, other nasal or palatal congenital anomalies, history of chronic exposure to allergens, or living in areas characterized by air pollution, being passive smokers since birth, presence of autoimmune disorders, serum 25-HVD >50 nmol/L and presence of clinically evident HVD.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement | 3 to 6 months
  The effect of vitamin D supplemental therapy on pediatric asthma severity as judged by the score of ISSAC questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No